CLINICAL TRIAL: NCT02143973
Title: An Open Label Extension Study of the Safety and Anti-Pruritic Efficacy of Nalbuphine HCl ER Tablets in Hemodialysis Patients With Uremic Pruritus
Brief Title: Open Label Extension Study of Nalbuphine HCl ER in Hemodialysis Patients With Uremic Pruritus
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Trevi Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TR02ext; 2013-005626-29 (EudraCT Number)
Record Dates: First submitted 2014-05-19; First posted 2014-05-21 (Estimated); Results first posted 2020-09-07 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2020-08

CONDITIONS: Uremic Pruritus; Pruritus
Keywords: Uremic; Pruritus; Itch; Chronic Itch; Nalbuphine
MeSH Terms: conditions — Pruritus | interventions — Nalbuphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- nalbuphine HCl ER (Experimental): nalbuphine HCl ER titrated from a dose of 30 mg QD to 120 BID for up to 3 weeks based on tolerability and efficacy, then maintained for an additional 21 weeks. Total duration of 24 weeks.
  Interventions: Drug: nalbuphine HCl ER

INTERVENTIONS:
Drug: nalbuphine HCl ER — nalbuphine HCl ER
  Other Names: nalbuphine

SUMMARY:
The primary objective of the study is to evaluate the overall safety of nalbuphine HCL ER tablets during a treatment period of up to 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subject completed participation in the TR02 study
* Subject is currently receiving in-center hemodialysis at the time of consent

Exclusion Criteria:

* Subject receiving or anticipated to be receiving nocturnal dialysis or home hemodialysis treatment during the study
* Subject received opiates on a daily basis during the 1 week prior to screening
* Other than the TR02 Study Drug, Subject received any investigational drug within 4 weeks prior to Screening
* Subject is a pregnant or lactating female

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2014-09; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Development Officer, Study Director — Trevi Therapeutics
Locations (35):
- United States (35):
  - Nephrology Associates PC, Birmingham, Alabama
  - University South Alabama Medical Center, Mobile, Alabama
  - Arizona Kidney Disease and Hypertension Center, Phoenix, Arizona
  - U.S. Renal Care Inc., Pine Bluff, Arkansas
  - North America Research Institute, Azusa, California
  - Pegasus Dialysis Center, Bakersfield, California
  - Central Nephrology Medical Group, Bakersfield, California
  - Mark Lee MD, Inc, Whittier, California
  - Nephrology and Hypertension Associates PC, Middlebury, Connecticut
  - Pines Clinical Research, Pembroke Pines, Florida
  - Genesis Clinical Research, Tampa, Florida
  - DaVita Central Orlando Dialysis, Winter Park, Florida
  - Southwest Georgia Nephrology Clinic PC, Albany, Georgia
  - Renal Physicians of Georgia, Macon, Georgia
  - Pacific Renal Research Institute, Meridian, Idaho
  - Fresenius Medical Care of Evergreen Park, Evergreen Park, Illinois
  - Western New England Renal and Transplant Association, Springfield, Massachusetts
  - Nephrology Center DBA Paragon Health, Kalamazoo, Michigan
  - McComb Limited Care Facility, McComb, Mississippi
  - Kidney Associates of Kansas City PC, Kansas City, Missouri
  - Nephrology-Hypertension Associates of Central New Jersey PA, North Brunswick, New Jersey
  - Renal Medicine Associates, Albuquerque, New Mexico
  - Newtown Dialysis Center Inc, Astoria, New York
  - Durham Nephrology Associates, Durham, North Carolina
  - Wake Nephrology Associates PA, Raleigh, North Carolina
  - Brookview Hills Research Associates LLC, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Nephrology Research Consortium, Bethlehem, Pennsylvania
  - Delaware Valley Nephrology, Philadelphia, Pennsylvania
  - Dialysis Clinic, Inc., Philadelphia, Pennsylvania
  - Carolina Diabetes and Kidney Center, Sumter, South Carolina
  - SouthEast Renal Research Institute, Chattanooga, Tennessee
  - U.S. Renal Care, Inc., Fort Worth, Texas
  - U.S. Renal Care Inc., Fort Worth, Texas
  - U.S. Renal Care Inc, Mansfield, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Nalbuphine HCl ER: nalbuphine HCl ER
  nalbuphine HCl ER BID: nalbuphine HCl ER titrated from 30 mg QD to 120 mg BID over three weeks based on tolerability and efficacy, then maintain dosing at that maximum achieved level; full titration and maintenance is 24 weeks.
Period: Overall Study
Arm/Group | Nalbuphine HCl ER
Started | 167
Completed | 101
Not Completed | 66

BASELINE CHARACTERISTICS:
Arm/Group | Nalbuphine HCl ER
Number analyzed (Participants) | 167
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.1 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75
  Male | 92
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31
  Not Hispanic or Latino | 136
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 89
  White | 73
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 146
  Europe | 21

OUTCOME MEASURES:

1. Primary Outcome: Number and Percetage of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: The number of participants reporting at least one TEAE of a particular body system and preferred term are reported (incidence)
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Nalbuphine HCl ER
Number analyzed (Participants) | 167
Participants | 133

ADVERSE EVENTS:
Arm/Group | Nalbuphine HCl ER
All-Cause Mortality (participants affected / at risk) | 0/167
Serious Adverse Events (participants affected / at risk) | 54/167
Other Adverse Events (participants affected / at risk) | 0/167
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nalbuphine HCl ER (N=167)
Arteriovenous graft site infection (Infections and infestations) | 4
Sepsis (Infections and infestations) | 3
Diverticulitis (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 2
Septic shock (Infections and infestations) | 2
Abcess neck (Infections and infestations) | 1
Arthritis bacterial (Infections and infestations) | 1
Bronchitis bacterial (Infections and infestations) | 1
Clostridium difficile infection (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Endometritis (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Urospesis (Infections and infestations) | 1
Syncope (Nervous system disorders) | 2
Ataxia (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 1
Haemorrhagic stroke (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Speech disorder (Nervous system disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Hypotension (Vascular disorders) | 3
Hypertension (Vascular disorders) | 2
Orthostatic hypotension (Vascular disorders) | 2
Hypertensive emergency (Vascular disorders) | 1
Jugular vein thrombosis (Vascular disorders) | 1
Malignant hypertension (Vascular disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Colitis (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal inflammation (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Proctitis (Gastrointestinal disorders) | 1
Retroperitoneal haematoma (Gastrointestinal disorders) | 1
Umbilical hernia (Gastrointestinal disorders) | 1
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1
Arteriovenous graft site hemorrhage (Injury, poisoning and procedural complications) | 1
Dialysis related complication (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1
Vascular graft complication (Injury, poisoning and procedural complications) | 1
Non-cardiac chest pain (General disorders) | 4
Sudden cardiac death (General disorders) | 1
Systemic inflammatory response syndrome (General disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Cardiac failure acute (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Fluid overload (Metabolism and nutrition disorders) | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 2
Cholangitis (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Anticoagulation drug level below therapeutic (Investigations) | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No